CLINICAL TRIAL: NCT04766229
Title: A Multimodal Technology-assisted Intervention for the Management of Menopause After Cancer: The Menopause After Cancer Study
Brief Title: The Menopause After Cancer Study
Acronym: MACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Irish Cancer Society (Other); Big Health Inc. (Industry); myPatientSpace (Unknown)
Responsible Party: Principal Investigator, Donal Brennan, Professor of Gynaecological Oncology, University College Dublin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RS21-002
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Menopause; Cancer; Insomnia
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): All participants in single arm study
  Interventions: Combination Product: Citalopram +/- Gabapentin + Sleepio + support person

INTERVENTIONS:
Combination Product: Citalopram +/- Gabapentin + Sleepio + support person — All participants will receive citalopram and/or gabapentin to manage vasomotor symptoms of menopause and will get access to digital CBT for insomnia and be asked to identify a support person

SUMMARY:
This study will recruit women with vasomotor symptoms of menopause and a prior cancer diagnosis, for whom conventional menopausal hormone therapy (MHT) is contraindicated for any reason. This study will examine if the addition of psycho-social support and digital cognitive behavioral therapy (CBT) for insomnia to standard non-hormonal pharmacotherapy can improve quality of life for these women.

DETAILED DESCRIPTION:
Patients who are eligible and provide informed consent will be enrolled into this single arm study. Patients will be prescribed non-hormonal pharmacotherapy tailored to the timing of their predominant symptoms. They will be given access to an evidence based platform for digital CBT for insomnia and asked to identify a partner or other companion who will commit to providing psychosocial support to the research participant throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Females over 18 years of age at the time of recruitment and onboarding.
2. Vasomotor symptoms of menopause
3. Previous or current cancer diagnosis
4. Conventional menopausal hormone therapy contraindicated for any reason
5. Can speak and read English proficiently
6. Competent using the internet and has access to smartphone or similar device

Exclusion Criteria:

1. ECOG performance status >3
2. Use of study medications to manage menopausal symptoms in the preceding 6 months
3. Use of CBT for insomnia in the preceding 6 months
4. Any contraindication to study medications
5. No internet access or competency issue with internet use
6. Unable to complete questionnaires or give informed consent
7. Current major mental illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Global Quality of Life scores as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30) instrument | 6 months
  Global quality of life will be assessed using the EORTC QLQ C30 questionnaire. This is a 30 item questionnaire which has been extensively validated internationally and is specific to patients treated for cancer. Minimum global quality of life score is 0 with a maximum of 100 with a higher score representing a better quality of life.

SECONDARY OUTCOMES:
Bother/Interference of vasomotor symptoms of menopause as measured by the Hot Flush Rating Scale | 6 months
  This will be measured by the Hot Flush Rating Scale which measures both frequency and impact of vasomotor symptoms. For this scale the minimum score is 1 and maximum score is 10 with higher scores indicating a greater degree of bother/interference.
Sleep dysfunction as measured by the Sleep Condition Indicator | 6 months
  This will be measured using the Sleep Condition Indicator tool. Minimum score is 0 with maximum score of 32 with higher scores indicating better sleep.

OTHER OUTCOMES:
Communication between participants and support person as measured by the Couples' Illness Communication Score. | 6 months
  Will be measured quantitatively using Couples' Illness Communication Score. The minimum score of 8 and a maximum score of 40 with higher scores indicating better communication.
The experience of participating in the couples communication aspect of the study | 6 months
  This will be explored qualitatively using semi structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Donal Brennan, PhD, Principal Investigator — UCD Dublin
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St. Vincent's University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers

REFERENCES:
- [Derived] Donohoe F, O'Meara Y, Roberts A, Comerford L, Kelly CM, Walshe JM, Peate M, Hickey M, Brennan DJ. The menopause after cancer study (MACS) - A multimodal technology assisted intervention for the management of menopausal symptoms after cancer - Trial protocol of a phase II study. Contemp Clin Trials Commun. 2021 Nov 11;24:100865. doi: 10.1016/j.conctc.2021.100865. eCollection 2021 Dec. PMID 34869938